CLINICAL TRIAL: NCT04220593
Title: Effects of Transcranial Direct Current Stimulation Associated With Cognitive Training in Alzheimer's Disease: Clinical Trials, Triple-blind and Randomized
Brief Title: Effects of Transcranial Direct Current Stimulation Associated With Cognitive Training in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, principal investigator and teacher, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CogAD
Record Dates: First submitted 2019-11-26; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- aETCC before TCog (Experimental): Anodic transcranial direct current stimulation (tDCS) over left dorsolateral prefrontal cortex (DLPFC) associated with cognitive training (Tcog). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Other: tDCS associated with Tcog
- aETCC during TCog (Experimental): Anodic transcranial direct current stimulation (tDCS) over left dorsolateral prefrontal cortex (DLPFC) associated with cognitive training (Tcog). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Other: tDCS associated with Tcog
- aETCC after TCog (Experimental): Anodic transcranial direct current stimulation (tDCS) over left dorsolateral prefrontal cortex (DLPFC) associated with cognitive training (Tcog). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Other: tDCS associated with Tcog
- Simulated aETCC during TCog (Sham Comparator): Anodic transcranial direct current stimulation (tDCS) over left dorsolateral prefrontal cortex (DLPFC) associated with cognitive training (Tcog). Duration: 20 minutes; Intensity: 2mA.
  Interventions: Other: tDCS associated with Tcog

INTERVENTIONS:
Other: tDCS associated with Tcog — 2mA-intensity aETCC will be applied to the left dorsolateral prefrontal cortex (CPFDL) region for 20 min, three times a week (every other day) over a one-month period, totaling 12 sessions. In each session activities aimed at stimulating cognition will be applied over the 20 minutes.

SUMMARY:
Alzheimer's disease (AD) is characterized by a progressive decline in cognitive functions, interfering with autonomy and independence. According to the Diagnostic and Statistical Manual of Mental Disorders (DSM 5), mnemonic dysfunction in AD must be related to aphasia, apraxia, agnosia, or changes in executive function. The clinical picture of the disease can be described as mild, moderate and severe. In the mild phase, the patient is disoriented and with difficulties in thinking, in later stages memory lapses become more intense and frequent. The symptoms of apraxia, aphasia and agnosia appear, causing a noticeable impact on the performance of simple daily activities, and neuropsychiatric and behavioral symptoms are expressed. Existing pharmacological treatments for AD treatment are able to minimize the symptoms of the disease, but are not able to promote cure. Therefore, studies have sought to better understand non-pharmacological strategies, aiming at optimizing the benefits of using the drug. Studies have suggested that tDCS promotes significant effects on cognitive processes assessed through cognitive tasks, not only in healthy individuals but also in clinical populations. Cognitive training (TCog) has similarly shown excellent results in the treatment of cognitive deficits due to AD. Thus, the present study aims to investigate when (before, during or after) the tDCS should be applied to potentiate the effects of TCog in people with AD by comparing four protocols of application of neurostimulation associated with TCog.

DETAILED DESCRIPTION:
It consists of a randomized, triple-blind, placebo-controlled clinical trial. The AETCC must be associated with the Tcog. Patients diagnosed in mild to moderate AD will be randomized into four groups: G1, aETCC before TCog; G2, aETCC during TCog; G3 aETCC after TCog and G4: simulated aETCC during TCog. Groups G1, G2 and G3 will receive the active current, while G4 will receive the simulated current. In each condition, an initial baseline assessment (T0) will be performed after 12 sessions (T1) and three weeks after the end of interventions (T2). The outcomes evaluated will be: cognition, executive function, functionality, neuropsychiatric symptoms and occupational performance. For all analyzes, SPSS (Statistical Package for Social Sciences - SPSS Inc, Chicago IL, USA) for Windows, Version 20.0, will be used and considered as significant, an alpha value of 5% (p <0.05 ).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study following the following requirements: (a) age between 55 and 85 years; (b) probable diagnosis AD; (c) scores higher than 18 on the Mini Mental State Examination (MMSE); (e) did not receive regular cognitive intervention within 3 months prior to the start of this clinical trial.

Exclusion Criteria:

* Patients will be excluded from this study while not meeting the following criteria: (a) individuals with severe metabolic and / or cardiac disorders, alcoholism, focal neurological disorders and associated psychiatric disorders; (b) use of hypnotics and benzodiazepines two weeks prior to study initiation; or (c) use of medication with cholinergic inhibitors and memantine for more than two months prior to this clinical trial; (d) or with any condition that could impair the neuropsychological assessment process or receive a cognitive intervention protocol from the study will be excluded from the study. In addition, participants with transient or definitive pacemakers, cochlear implants, or intracranial aneurysm clips will be excluded; (e) individuals with a history of seizures; (f) the presence of tumors, epilepsy or substance abuse.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive function by the Alzheimer's Disease Assessment Scale (ADAS-Cog) | baseline, after 4 weeks and after 12 weeks
  Cognitive Scale of the Alzheimer's Disease Assessment Scale (ADAS-Cog), consisting of 11 items that assesses performance related to memory, language, praxis and comprehension skills, with a maximum score of 70 points. Thus, the higher the score, the more compromised the individual is. Application takes about 30 minutes (Mohs & Cohen, 1988). In addition, the Montreal Cognitive Assessment (MoCA), a cognitive screening tool created by Nasreddine et al. (2005).
Change in global cognitive function by the Montreal Cognitive Assessment (MoCA) | baseline, after 4 weeks and after 12 weeks
  MoCA is composed of eight cognitive domains, which are scored within a range of 0 to 30 points (higher scores indicate better function): short-term memory; visuospatial skills; executive function; verbal fluency; attention, concentration and working memory; language; sentence repetition; and spatiotemporal orientation.

SECONDARY OUTCOMES:
Change in Executive Function by the Trail Making Test (TMT) | baseline, after 4 weeks and after 12 weeks
  The Trail Making Test (TMT) will be administered (Reitan, 1958). From a clinical point of view, TMT is widely used as an indicator of brain dysfunction. TMT is divided into two parts, TMT-A and TMT-B. In the first, circles numbered 1 to 25 following the randomly arranged numerical sequence should be connected, time taken and considered, ie the task should be performed as soon as possible. In the TMT-B task, the connection must alternate between numbers and letters. The TMT (AB) scores consist of the time taken to complete each part, other derived scores are used, such as the difference score (TMT-B - TMT-A) and the ratio score (TMT-A) / TMT- B) (Llinàs-Reglà et al, 2015).
Change in Executive Function by the Tower of London | baseline, after 4 weeks and after 12 weeks
  The Tower of London (Shallice, 1982) has been used in studies to evaluate executive function in elderly with AD (Satler, Guimarães, Tomaz, 2016). Tower of London is made up of three vertical pins of different heights and three colored spheres, with a hole in the center to fit the pins. The goal is to move them to reproduce, in a given number of moves, the position of a presented target figure. There are 15 problems with increasing difficulty and reduced possibilities for moving parts. Three attempts to resolve the issue are allowed. Will be evaluated: total and average execution time, and total score, obtained by the sum of the points of each step, ranging from 0 to 3.
Change in Functionality by the Disability Assessment for Dementia (DAD) | baseline, after 4 weeks and after 12 weeks
  Disability Assessment for Dementia (DAD) (Gauthier, et al., 1997; Gélinas et al., 1999). The DAD comprises 17 items that assess ADLs and 23 items that assess instrumental ADL (iADL) and leisure activities. In the category related to ADLs are evaluated hygiene, dressing, undressing, continence and food. IADL assessment and leisure activities consist of tasks related to meal preparation, phoning, sightseeing, finances and correspondence, medication and leisure, and housework (Feldman et al. (2001; Suh et al., 2004). maximum score is 100, lower scores indicate higher level of impairment (Bahia et al., 2010).
Change in Neuropsychiatric symptoms by the Neuropsychiatric Inventory Questionnaire (NPI-Q) | baseline, after 4 weeks and after 12 weeks
  This outcome will be assessed with the Neuropsychiatric Inventory Questionnaire (NPI-Q; Kaufer et al., 2000). This instrument consists of a self-administered caregiver scale and provides information on 12 characteristic behavioral and psychological symptoms in patients with dementia. The severity level will be identified (1 = mild, 2 = moderate, 3 = severe). The overall severity score ranges from 0 to 36, with zero indicating no neuropsychiatric symptoms. The reliability and validity of this modified NPI score have been previously established (NPI-Q; Kaufer et al., 2000).
Change in Occupational performance by theCanadian Occupational Performance Measure (COPM) | baseline, after 4 weeks and after 12 weeks
  The Canadian Occupational Performance Measure (COPM) (Law et al., 2009) will be used to assess occupational performance, ie engagement in daily activities. The COPM is can be applied with the patient or caregiver, following four steps, firstly it seeks to identify which areas of occupational performance are impaired, ie, which occupations are compromised, and then assign a value from 1 to 10 to measure the degree of importance that the activities listed have for the interviewee or caregiver. Next, five of these activities are organized by priority, and each of them should be assigned a value between 1 and 10 to describe the interviewee's performance and satisfaction respectively. In the end, the averages of performance and satisfaction are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Universidade Federal da Paraíba
Locations (1):
- Suellen Andrade, João Pessoa, Paraíba, Brazil